CLINICAL TRIAL: NCT01723501
Title: Whole Body Cleansing With 0.25% Chlorhexidine at Birth for Prevention of Sepsis in Infants <1500 g: a Multi-center, Blinded, Randomized Trial
Brief Title: Chlorhexidine Skin Application for Prevention of Infection in Infants Weighing <1500 g at Birth
Acronym: CAPS
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was not started and prematurely closed.
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Maulana Azad Medical College (Other); Vardhman Mahavir Medical College And Safdarjung Hospital (Other)
Responsible Party: Principal Investigator, Dr Vinod K Paul, Professor & Head, Department of Pediatrics, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NHKC-Chx2012
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Neonatal Sepsis; Neonatal Mortality Rate
Keywords: chlorhexidine; sepsis; neonatal; whole-body skin cleansing
MeSH Terms: conditions — Neonatal Sepsis; Sepsis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sterile water (Placebo Comparator): sterile water wipes
  Interventions: Drug: sterile water
- 0.25% chlorhexidine (Experimental): 0.44% chlorhexidine digluconate wipes which will release 0.25% free chlorhexidine
  Interventions: Drug: 0.25% chlorhexidine

INTERVENTIONS:
Drug: 0.25% chlorhexidine — 0.44% chlorhexidine di-gluconate body wipes which would release 0.25% free chlorhexidine on application
  Other Names: Chx
  Arms: 0.25% chlorhexidine
Drug: sterile water — Sterile water wipes (placebo)
  Arms: sterile water

SUMMARY:
Purpose of this study is determine if skin application of chlorhexidine at birth would reduce infection in infants weighing <1500 g at birth.

DETAILED DESCRIPTION:
Background

Infants weighing <1500 g at birth infants are more prone to acquire infections, often through their immature skin which serve as a portal of entry for invasive pathogens. Skin application of antiseptics such as chlorhexidine may reduce infections in these infants. However, there is a paucity of data on the safety and efficacy of such intervention in these infants.

Hypothesis:

Among hospitalized very low birth weight (VLBW; <1500 g) neonates, single whole body skin cleansing with 0.25% chlorhexidine within 6 hours after birth would reduce the incidence of sepsis in the first seven days of life from 25% to 17.5% (relative reduction of 30%) when compared to skin cleansing with sterile water

Objectives:

Primary- To evaluate the effect of whole body skin cleansing with 0.25% chlorhexidine (single application, at birth) on the incidence of sepsis (culture positive or culture negative) compared to sterile water cleansing in the first week of life in VLBW infants

Secondary- to compare following outcomes in this experiment:

1. Culture-confirmed sepsis within the first week of life
2. Need for repeat hospital admissions within first 28 days of life
3. Mortality within first 28 days of life
4. Cold stress/hypothermia at 0, 5, 15 and 30 minutes of intervention
5. Skin condition at 24 h of life
6. Colonization rates (subset)
7. Serum levels of chlorhexidine (subset)

Methods:

Eligible infants would be randomized within 6 hours of birth to either whole body skin cleansing with chlorhexidine (specially prepared wipes releasing 0.25% chlorhexidine), or sterile water (placebo). The research staff would collect the baseline data, record the axillary temperature and assess the skin condition using the Newborn Skin Condition Scoring (NSCS)score. The research team would follow the infants for development of sepsis and other outcomes. The infants would be subjected to detailed sepsis work up on clinical suspicion of sepsis, until 28 days of life.

Sepsis would be defined based on combination of clinical course, indirect markers, bacterial culture results and antibiotic treatment status.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight less than 1500 g

Exclusion Criteria:

* Birth weight <750 g
* Major congenital malformations
* Total duration of positive pressure ventilation (PPV) > 3 mins OR chest compressions
* Shock- requiring inotropes >10 mic/kg/min

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-11

PRIMARY OUTCOMES:
Sepsis within first 7 days of life | First 7 days of life
  Sepsis would be defined on the basis of clinical course, lab parameters including culture results and antibiotic treatment given.

SECONDARY OUTCOMES:
Readmissions & mortality rates within neonatal period | 28 days
  The re-admissions & mortality rates within neonatal period in these infants will be prospectively recorded during hospital admission as well as follow up. The follow up includes telephonic contact as well as home visits and verbal autopsy in cases of deaths at home.
Body temperature at 0, 5, 15, 30 minutes after application | 30 minutes
  Axillary temperature would be monitored with thermometer at above time points for full three minutes.
Skin condition | 24 ±6 hours
  Newborn Skin Condition Score (NSCS)will be used to assess the skin condition.
Skin colonization rates | 24 ±6 hours
  In a sub-group of infants, skin swabs will be collected at baseline and 24 ±6 hours and sent to microbiology lab; colonization rates would be determined by semi-quantitative methods.
Chlorhexidine percutaneous absorption | 48 ±6 hours
  Serum chlorhexidine levels will be assayed in a sub-set to assess the extent of percutaneous absorption. 5ml of blood will be stored at -80 deg. C till transport to the lab. Samples will be processed in batches as per standard protocol to determine the levels.

CONTACTS AND LOCATIONS:
Overall Officials: Vinod K Paul, MD, PhD, Principal Investigator — All India Institute of Medical Sciences
Locations (3):
- India (3):
  - Maulana Azad Medical College, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Vardhman Medical College and Safdarjung Hospital, New Delhi, National Capital Territory of Delhi

REFERENCES:
- See also: Related Info — http://www.newbornwhocc.org